CLINICAL TRIAL: NCT05807113
Title: Assessment of Skin Tolerance and Efficacy of a Cosmetic Product After 5 Days of Use on Subjects With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CS02AC-ICBD
Record Dates: First submitted 2023-02-15; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-02

CONDITIONS: Atopic Diathesis; Eczema-prone Skin

STUDY DESIGN:
Intervention Model Description: intra-individual comparison
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atopi intensive care BNO 3731 for topical use (Experimental)
  Interventions: Other: Atopi intensive care BNO 3731
- Benchmark skin care product for topical use (Active Comparator)
  Interventions: Other: Benchmark product

INTERVENTIONS:
Other: Atopi intensive care BNO 3731 — Crem twice daily
  Arms: Atopi intensive care BNO 3731 for topical use
Other: Benchmark product — Crem twice daily
  Arms: Benchmark skin care product for topical use

SUMMARY:
The aim of this study is to compare the efficacy and tolerability and of a cosmetic product to one that is already available on the market (benchmark product). Efficacy is assessed by instrumental measurements of skin condition, clinical examinations, and questionnaires.

DETAILED DESCRIPTION:
The objective of this exploratory study is to investigate the efficacy and tolerability of a cosmetic product on subjects with atopic dermatitis after 5 days of use in comparison to a benchmark product.

The efficacy will be evaluated via instrumental measurements of skin hydration by Corneometer, transepidermal water loss by Tewameter and erythema by Chromameter as well as by evaluation of itch by using a Numerical Rating Scale (NRS). For efficacy and tolerability evaluation an objective and, in the case of adults, an additional subjective dermatological assessment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent of the subject to participate in the study, or, for underaged subjects of the parents/ legal guardians to let their child participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits or, for underaged subjects, willingness of the parents/ legal guardians to actively support their child's participation in the study and to come to the scheduled visits with their child
* Female and/or male
* Children from 6 months to 14 years of age and Adult subjects between 18 and 65 years of age
* Eczema-prone skin and atopic diathesis, diagnosed by the dermatologist

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* Insulin-dependent diabetes mellitus
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension, cardiovascular diseases
* Documented allergies to cosmetic products and/ or ingredients, skin care and/or skin cleansing products
* Wounds, moles, tattoos, scars, excessive hair growth, etc. at the test area that could influence the investigation
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids) and/or antihistamines (e.g. antiallergics) within the last 7 days prior to the start of the study
* Systemic therapy with anti-phlogistic agents or analgetics (e.g. diclophenac), except for minor pain relief medicine like acetylsalicylic acid or paracetamol within the last 3 days prior to the start of the study

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in transepidermal water loss (g/m2h) | after 6 days of treatment
Mean change from baseline in skin redness by Chromameter | after 6 days of treatment
Mean change from baseline in skin hydration (Skin capacitance by Corneometer [a.u.]) | after 6 days of treatment
Changes from baseline in objective dermatological evaluation of skin status (erythema, dryness, scaling, fissures, papules, pustules, edema, vesicles, weeping) by dermatologist (min=0, max=3; 3=worse outcome) | after 6 days of treatment

SECONDARY OUTCOMES:
Change from baseline in the scoring of subjective dermatological evaluation via questionnaire (adults) (min=0, max=3; 3=worse outcome) | after 6 days of treatment
Subjective evaluation of itch on Numeric Rating Scale (NRS-11) (min= 0, max=10, 10 = worst imaginable itch) | every day, day 1 until 6 days of treatment
Evaluation of products traits via questionnaire (20 questions with different answers, no scales) | after 6 days of treatment
Safety of BNO 3732 measured by reported Adverse Events | until day 29

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Laing, Dr., Principal Investigator — proDERM GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Germany